CLINICAL TRIAL: NCT03400332
Title: A Phase 1/2 Study of BMS-986253 in Combination With Nivolumab or Nivolumab Plus Ipilimumab in Advanced Cancers
Brief Title: A Study of BMS-986253 in Combination With Nivolumab or Nivolumab Plus Ipilimumab in Advanced Cancers
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CA027-002; 2023-509061-20 (Registry Identifier: EU Trial Number)
Record Dates: First submitted 2018-01-12; First posted 2018-01-17 (Actual); Results first posted 2025-06-19 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Cancer; Melanoma
MeSH Terms: conditions — Neoplasms; Melanoma | interventions — HuMax-IL8; Nivolumab; Ipilimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part 1A: BMS-986253 + nivolumab (Experimental)
  Interventions: Drug: BMS-986253; Biological: Nivolumab
- Part 1B: BMS-986253 + nivolumab (Experimental)
  Interventions: Drug: BMS-986253; Biological: Nivolumab
- Part 1C: BMS-986253 + nivolumab + ipilimumab (Experimental)
  Interventions: Drug: BMS-986253; Biological: Nivolumab; Biological: Ipilimumab
- Part 2A: BMS-986253 + nivolumab + ipilimumab (Experimental)
  Interventions: Drug: BMS-986253; Biological: Nivolumab; Biological: Ipilimumab
- Part 2B: Placebo + nivolumab + ipilimumab (Placebo Comparator)
  Interventions: Biological: Nivolumab; Biological: Ipilimumab; Other: Placebo

INTERVENTIONS:
Drug: BMS-986253 — Specified dose on specified days
  Arms: Part 1A: BMS-986253 + nivolumab; Part 1B: BMS-986253 + nivolumab; Part 1C: BMS-986253 + nivolumab + ipilimumab; Part 2A: BMS-986253 + nivolumab + ipilimumab
Biological: Nivolumab — Specified dose on specified days
  Other Names: BMS-936558; Opdivo
Biological: Ipilimumab — Specified dose on specified days
  Other Names: BMS-734016; YERVOY
  Arms: Part 1C: BMS-986253 + nivolumab + ipilimumab; Part 2A: BMS-986253 + nivolumab + ipilimumab; Part 2B: Placebo + nivolumab + ipilimumab
Other: Placebo — Specified dose on specified days
  Arms: Part 2B: Placebo + nivolumab + ipilimumab

SUMMARY:
The purpose of this study is to investigate experimental medication BMS-986253 in combination with Nivolumab or Nivolumab plus Ipilimumab in participants with advanced cancers.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic confirmation of a solid tumor that is advanced (metastatic, recurrent and/or unresectable) with measurable disease per RECIST v1.1
* At least 1 lesion accessible for biopsy
* Eastern Cooperative Oncology Group Performance Status of 0 or 1

Exclusion Criteria:

* Participants with CNS metastases as the only site of active disease (Participants with controlled brain metastases; however, will be allowed to enroll)
* Participants with active, known or suspected autoimmune disease
* Participants with conditions requiring systemic treatment with either corticosteroids (> 10mg prednisone equivalents) or other immunosuppressive medications within 14 days of study treatment administration
* Participants with a known history of testing positive for Human Immunodeficiency Virus (HIV) or known Acquired Immunodeficiency Syndrome (AIDS)
* Cytotoxic agents, unless at least 4 weeks have elapsed from last dose of prior anti-cancer therapy and initiation of study therapy

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 281 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2024-04-26 (Actual); Study Completion 2025-11-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (72):
- United States (29):
  - Local Institution - 0059, Springdale, Arkansas
  - Local Institution - 0099, Los Angeles, California
  - Local Institution - 0007, Lakewood, Colorado
  - Local Institution - 0087, Atlanta, Georgia
  - Local Institution - 0100, Atlanta, Georgia
  - Local Institution - 0101, Marietta, Georgia
  - Local Institution - 0012, Columbia, Maryland
  - Local Institution - 0003, Lutherville, Maryland
  - Local Institution - 0060, Boston, Massachusetts
  - Local Institution - 0004, Ann Arbor, Michigan
  - Local Institution - 0076, Omaha, Nebraska
  - Comprehensive Cancer Centers Of Nevada, Las Vegas, Nevada
  - Local Institution - 0005, Hackensack, New Jersey
  - Local Institution - 0032, New Brunswick, New Jersey
  - Local Institution - 0025, New York, New York
  - Local Institution - 0002, New York, New York
  - Local Institution - 0028, Oklahoma City, Oklahoma
  - Local Institution - 0017, Eugene, Oregon
  - Local Institution - 0001, Pittsburgh, Pennsylvania
  - Local Institution - 0009, Greenville, South Carolina
  - Local Institution - 0011, Austin, Texas
  - Local Institution - 0010, Dallas, Texas
  - Local Institution - 0014, Fort Worth, Texas
  - Local Institution - 0018, Houston, Texas
  - Local Institution - 0006, San Antonio, Texas
  - Local Institution - 0013, Tyler, Texas
  - Local Institution - 0058, Salt Lake City, Utah
  - Local Institution - 0015, Fairfax, Virginia
  - Local Institution - 0008, Norfolk, Virginia
- Australia (6):
  - Local Institution - 0088, Wollstonecraft, New South Wales
  - Local Institution - 0096, Adelaide, South Australia
  - Local Institution - 0090, Melbourne, Victoria
  - Local Institution - 0095, Melbourne, Victoria
  - Local Institution - 0097, Perth, Western Australia
  - Local Institution - 0091, Ballarat Central
- Belgium (3):
  - Local Institution - 0037, Brussels
  - Local Institution - 0036, Ghent
  - Local Institution - 0082, Kortrijk
- Canada (6):
  - Local Institution - 0030, Edmonton, Alberta
  - Local Institution - 0029, Vancouver, British Columbia
  - Local Institution - 0078, Victoria, British Columbia
  - Local Institution - 0020, Toronto, Ontario
  - Local Institution - 0055, Toronto, Ontario
  - Local Institution - 0056, Montreal, Quebec
- France (5):
  - Local Institution - 0067, Marseille, Bouches-du-Rhône
  - Local Institution - 0085, Nantes
  - Local Institution - 0068, Paris
  - Local Institution - 0102, Toulouse
  - Local Institution - 0069, Villejuif
- Germany (4):
  - Local Institution - 0054, Tübingen, Baden-Wurttemberg
  - Local Institution - 0052, Mainz, Rhineland-Palatinate
  - Local Institution - 0034, Berlin
  - Local Institution - 0053, Hamburg
- Italy (4):
  - Local Institution - 0043, Forlì
  - Local Institution - 0042, Milan
  - Local Institution - 0027, Napoli
  - Local Institution - 0026, Rozzano-milano
- Poland (2):
  - Local Institution - 0071, Krakow
  - Local Institution - 0077, Warsaw
- Spain (6):
  - Local Institution - 0045, Madrid
  - Local Institution - 0022, Madrid
  - Local Institution - 0023, Madrid
  - Local Institution - 0044, Málaga
  - Local Institution - 0021, Pamplona
  - Local Institution - 0047, Santiago de Compostela
- Local Institution - 0049, Lund, Sweden
- Switzerland (3):
  - Local Institution - 0040, Lausanne
  - Local Institution - 0041, Sankt Gallen
  - Local Institution - 0039, Zurich
- United Kingdom (3):
  - Local Institution - 0024, Manchester, Greater Manchester
  - Local Institution - 0083, Glasgow, Lanarkshire
  - Local Institution - 0019, Birmingham, West Midlands

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 281 participants were randomized and 278 received treatment.
  Part 1: 159 participants were directly treated and not blinded (open label).
  Part 2: 122 participants were double-blinded and randomized. 122 participants were randomized in the pre-treatment phase while 119 received treatment. 3 participants were randomized but did not receive treatment.
Groups:
- Part 1: 600 Q4W: 600 mg BMS-986253 Q4W + 480 mg nivolumab Q4W
- Part 1: 1200 Q4W: 1200 mg BMS-986253 Q4W + 480 mg nivolumab Q4W
- Part 1: 2400 Q4W: 2400 mg BMS-986253 Q4W + 480 mg nivolumab Q4W
- Part 1: 1200 Q2W: 1200 mg BMS-986253 Q2W + 480 mg nivolumab Q4W
- Part 1: 2400 Q2W: 2400 mg BMS-986253 Q2W + 480 mg nivolumab Q4W
- Part 1: 3600 Q2W: 3600 mg BMS-986253 Q2W + 480 mg nivolumab Q4W
- Part 1: 3600Q2W + Nivo + Ipi: 3600 mg BMS-986253 Q2W + nivolumab 1 mg/kg Q3W (480 mg Q4W after 12 Weeks) + ipilimumab 3 mg/kg Q3W
- Part 2 Arm A: BMS+Nivo+Ipi: BMS-986253 3600 mg Q2W + nivolumab 1 mg/kg Q3W + ipilimumab 3 mg/kg Q3W for 12 weeks; BMS-986253 3600 mg Q2W + nivolumab 480 mg Q4W thereafter
- Part 2 Arm B: Placebo+Nivo+Ipi: Placebo Q2W + nivolumab 1 mg/kg Q3W + ipilimumab 3 mg/kg Q3W for 12 weeks; BMS-986253 3600 mg Q2W + nivolumab 480 mg Q4W thereafter
Period: Pre-Treatment
Arm/Group | Part 1: 600 Q4W | Part 1: 1200 Q4W | Part 1: 2400 Q4W | Part 1: 1200 Q2W | Part 1: 2400 Q2W | Part 1: 3600 Q2W | Part 1: 3600Q2W + Nivo + Ipi | Part 2 Arm A: BMS+Nivo+Ipi | Part 2 Arm B: Placebo+Nivo+Ipi
Started | 16 | 15 | 18 | 12 | 63 | 20 | 15 | 62 | 60
Randomized | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 62 | 60
Completed (Treated) | 16 | 15 | 18 | 12 | 63 | 20 | 15 | 62 | 57
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Not completed — Other reasons | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — No longer met study criteria | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Period: Treatment
Arm/Group | Part 1: 600 Q4W | Part 1: 1200 Q4W | Part 1: 2400 Q4W | Part 1: 1200 Q2W | Part 1: 2400 Q2W | Part 1: 3600 Q2W | Part 1: 3600Q2W + Nivo + Ipi | Part 2 Arm A: BMS+Nivo+Ipi | Part 2 Arm B: Placebo+Nivo+Ipi
Started (Started=Received study treatment) | 16 | 15 | 18 | 12 | 63 | 20 | 15 | 62 | 57
Completed (Completed=continuing in study) | 11 | 10 | 15 | 9 | 51 | 14 | 11 | 58 | 49
Not Completed | 5 | 5 | 3 | 3 | 12 | 6 | 4 | 4 | 8
Not completed — Participant withdrew consent | 2 | 2 | 0 | 0 | 3 | 3 | 1 | 1 | 1
Not completed — Other reasons | 0 | 1 | 1 | 0 | 3 | 1 | 2 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 3 | 1 | 2 | 3 | 6 | 2 | 1 | 3 | 6

BASELINE CHARACTERISTICS:
Population: All treated participants for Part 1 and all randomized participants for Part 2. Participants in Part 1 were not randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: 600 Q4W | Part 1: 1200 Q4W | Part 1: 2400 Q4W | Part 1: 1200 Q2W | Part 1: 2400 Q2W | Part 1: 3600 Q2W | Part 1: 3600Q2W + Nivo + Ipi | Part 2 Arm A: BMS+Nivo+Ipi | Part 2 Arm B: Placebo+Nivo+Ipi | Total
Number analyzed (Participants) | 16 | 15 | 18 | 12 | 63 | 20 | 15 | 62 | 60 | 281
Age, Continuous [Mean (Full Range); unit: Years] | 60.4 [35.0 to 86.0] | 64.6 [49.0 to 83.0] | 66.3 [40.0 to 82.0] | 64.4 [51.0 to 87.0] | 63.0 [43.0 to 86.0] | 62.6 [36.0 to 78.0] | 56.6 [32.0 to 79.0] | 62.3 [22.0 to 89.0] | 60.6 [22.0 to 83.0] | 62.2 [22.0 to 89.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 5 | 5 | 18 | 7 | 5 | 22 | 17 | 88
  Male | 11 | 11 | 13 | 7 | 45 | 13 | 10 | 40 | 43 | 193
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 1 | 0 | 4 | 0 | 0 | 0 | 1 | 8
  Not Hispanic or Latino | 16 | 13 | 17 | 9 | 40 | 13 | 10 | 42 | 41 | 201
  Unknown or Not Reported | 0 | 0 | 0 | 3 | 19 | 7 | 5 | 20 | 18 | 72
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 7
  White | 15 | 13 | 18 | 11 | 59 | 18 | 13 | 56 | 53 | 256
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 6 | 6 | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Adverse Events (AEs) - Part 1
Description: An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a pre-existing medical condition in a clinical investigation participant administered study treatment and that does not necessarily have a causal relationship with this treatment. Adverse events are graded on a scale from 1 to 5, with Grade 1 being mild and asymptomatic; Grade 2 is moderate requiring minimal, local or noninvasive intervention; Grade 3 is severe or medically significant but not immediately life-threatening; Grade 4 events are usually severe enough to require hospitalization; Grade 5 events are fatal.
  This endpoint was prespecified in the protocol to include only participants in Part 1.
Time Frame: From first dose up to 100 days after last dose (up to 65 months)
Population: All treated participants in Part 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: 600 Q4W | Part 1: 1200 Q4W | Part 1: 2400 Q4W | Part 1: 1200 Q2W | Part 1: 2400 Q2W | Part 1: 3600 Q2W | Part 1: 3600Q2W + Nivo + Ipi
Number analyzed (Participants) | 16 | 15 | 18 | 12 | 63 | 20 | 15
Participants | 16 | 14 | 18 | 12 | 60 | 20 | 15

2. Primary Outcome: Number of Participants Experiencing Serious Adverse Events (SAEs) - Part 1
Description: A serious adverse event is defined as any untoward medical occurrence that, at any dose: results in death, is life-threatening, requires inpatient hospitalization or causes prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is an important medical event.
  This endpoint was prespecified in the protocol to include only participants in Part 1.
Time Frame: From first dose up to 100 days after last dose (up to 65 months)
Population: All treated participants in Part 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: 600 Q4W | Part 1: 1200 Q4W | Part 1: 2400 Q4W | Part 1: 1200 Q2W | Part 1: 2400 Q2W | Part 1: 3600 Q2W | Part 1: 3600Q2W + Nivo + Ipi
Number analyzed (Participants) | 16 | 15 | 18 | 12 | 63 | 20 | 15
Participants | 13 | 10 | 13 | 7 | 31 | 12 | 9

3. Primary Outcome: Number of Participants Experiencing Dose Limiting Toxicities (DLTs) - Part 1
Description: Dose-Limiting Toxicities (DLTs) are effects of a treatment that are serious enough to prevent an increase in dose of that treatment, as advised by the Dose Review Team. DLTs will be defined based on the incidence, intensity, and duration of AEs that are possibly related to study treatment. DLTs will include gastrointestinal, hepatic, hematologic, dermatologic, and other AEs.
  This endpoint was prespecified in the protocol to include only participants in Part 1.
Time Frame: From first dose up to 100 days after last dose (up to 65 months)
Population: All treated participants in Part 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: 600 Q4W | Part 1: 1200 Q4W | Part 1: 2400 Q4W | Part 1: 1200 Q2W | Part 1: 2400 Q2W | Part 1: 3600 Q2W | Part 1: 3600Q2W + Nivo + Ipi
Number analyzed (Participants) | 16 | 15 | 18 | 12 | 63 | 20 | 15
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants Experiencing Adverse Events (AEs) Leading to Discontinuation - Part 1
Description: Number of participants with any grade adverse events (AEs) leading to discontinuation of study treatment. An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a pre-existing medical condition in a clinical investigation participant administered study drug and that does not necessarily have a causal relationship with this treatment. Toxicities will be graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.
  This endpoint was prespecified in the protocol to include only participants in Part 1.
Time Frame: From first dose up to 100 days after last dose (up to 65 months)
Population: All treated participants in Part 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: 600 Q4W | Part 1: 1200 Q4W | Part 1: 2400 Q4W | Part 1: 1200 Q2W | Part 1: 2400 Q2W | Part 1: 3600 Q2W | Part 1: 3600Q2W + Nivo + Ipi
Number analyzed (Participants) | 16 | 15 | 18 | 12 | 63 | 20 | 15
Participants | 3 | 2 | 3 | 3 | 7 | 1 | 3

5. Primary Outcome: Number of Participants Who Died - Part 1
Description: The number of participants who died due to any cause are summarized. This endpoint was prespecified in the protocol to include only participants in Part 1.
Time Frame: From first dose up to 100 days after last dose (up to 65 months)
Population: All treated participants in Part 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: 600 Q4W | Part 1: 1200 Q4W | Part 1: 2400 Q4W | Part 1: 1200 Q2W | Part 1: 2400 Q2W | Part 1: 3600 Q2W | Part 1: 3600Q2W + Nivo + Ipi
Number analyzed (Participants) | 16 | 15 | 18 | 12 | 63 | 20 | 15
Participants | 14 | 15 | 17 | 10 | 53 | 13 | 8

6. Primary Outcome: Most Frequently Reported Grade 3 and Grade 4 Laboratory Test Results - Part 1
Description: Laboratory results were graded using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Laboratory tests are graded on a scale from 1 to 5, with Grade 1 being mild and asymptomatic; Grade 2 is moderate requiring minimal, local or noninvasive intervention; Grade 3 is severe or medically significant but not immediately life-threatening; Grade 4 events are usually severe enough to require hospitalization; Grade 5 events are fatal.
  This endpoint was prespecified in the protocol to include only participants in Part 1.
Time Frame: From first dose up to 30 days after last dose (up to 63 months)
Population: All treated participants in Part 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: 600 Q4W | Part 1: 1200 Q4W | Part 1: 2400 Q4W | Part 1: 1200 Q2W | Part 1: 2400 Q2W | Part 1: 3600 Q2W | Part 1: 3600Q2W + Nivo + Ipi
Number analyzed (Participants) | 16 | 15 | 18 | 12 | 63 | 20 | 15
Participants
  Hemoglobin - Grade 3 | 2 | 1 | 2 | 2 | 7 | 3 | 3
  Alanine aminotransferase - Grade 3 | 0 | 1 | 0 | 0 | 0 | 0 | 2
  Alkaline phosphatase - Grade 3 | 0 | 0 | 2 | 0 | 2 | 3 | 2
  Aspartate aminotransferase - Grade 3 | 0 | 1 | 0 | 0 | 0 | 2 | 1
  Phosphate - Grade 3 | 0 | 1 | 2 | 0 | 3 | 1 | 0
  Sodium - Grade 3 | 0 | 2 | 1 | 0 | 5 | 1 | 2
  Lipase - Grade 3 | 1 | 1 | 2 | 1 | 3 | 0 | 2
  Lipase - Grade 4 | 0 | 0 | 0 | 1 | 2 | 0 | 2
  Amylase - Grade 3 | 0 | 0 | 1 | 0 | 0 | 0 | 2
  Amylase - Grade 4 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Albumin - Grade 3 | 0 | 0 | 3 | 0 | 2 | 0 | 0

7. Secondary Outcome: Objective Response Rate (ORR) - Part 1
Description: Objective Response Rate per investigator is the percentage of participants who have a confirmed complete or partial best overall response (BOR) among participants who have measurable disease at baseline. Complete Response (CR) is defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to =< 10 mm. Partial Response (PR) is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Baseline was defined as evaluations or events that occur before the date and time of the first dose of study treatment or evaluations on the same date and time of the first dose of study treatment were also considered as baseline evaluations. This endpoint was prespecified in the protocol to include only participants in Part 1.
Time Frame: From the date of the first dose to the date of first objectively documented progression per RECIST v1.1 or the date of subsequent therapy, whichever occurred first (up to approximately 74 months)
Population: All treated participants in Part 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part 1: 600 Q4W | Part 1: 1200 Q4W | Part 1: 2400 Q4W | Part 1: 1200 Q2W | Part 1: 2400 Q2W | Part 1: 3600 Q2W | Part 1: 3600Q2W + Nivo + Ipi
Number analyzed (Participants) | 16 | 15 | 18 | 12 | 63 | 20 | 15
Percentage of Participants | 6.3 [0.2 to 30.2] | 6.7 [0.2 to 31.9] | 16.7 [3.6 to 41.4] | 0 [0.0 to 26.5] | 3.2 [0.4 to 11.0] | 10.0 [1.2 to 31.7] | 13.3 [1.7 to 40.5]

8. Secondary Outcome: Duration of Response (DOR) - Part 1
Description: DOR for a participant with a best overall response (BOR) of CR or PR is defined as the date of first response up to the date of the first objectively documented tumor progression by the investigator per RECIST v1.1 or death, whichever occurs first. Analysis computed using Kaplan-Meier method.
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to =< 10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum during the study (this includes the baseline sum if that is the smallest on study). The sum must also demonstrate an absolute increase of at least 5 mm.
  This endpoint was prespecified in the protocol to include only participants in Part 1.
Time Frame: as for outcome 7
Population: All confirmed responders in Part 1
Measure: Median (Full Range); unit: Months
Arm/Group | Part 1: 600 Q4W | Part 1: 1200 Q4W | Part 1: 2400 Q4W | Part 1: 1200 Q2W | Part 1: 2400 Q2W | Part 1: 3600 Q2W | Part 1: 3600Q2W + Nivo + Ipi
Number analyzed (Participants) | 1 | 1 | 3 | 0 | 2 | 2 | 2
Months | 3.7 [3.7 to 3.7] | 28.9 [28.9 to 28.9] | 44.6 [8.4 to 44.6] |  | 21.09 [4.0 to 21.1] | 3.4 [3.4 to 3.4] | NA [3.7 to 24.0] — Median not calculated due to insufficient number of events

9. Secondary Outcome: Maximum Concentration (Cmax) - Part 1
Description: Cmax is the maximum (or peak) serum concentration that a drug achieves in a specified compartment or test area of the body after the drug has been administered and before the administration of a second dose.
  1 cycle=28 days for all Arms/Groups except in "Part 1: 3600Q2W + Nivo + Ipi" Arm/Group (1 cycle=42 days)
Time Frame: Cycle 1 Day 1
Population: All treated participants in Part 1 who have evaluable concentration-time data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Part 1: 600 Q4W | Part 1: 1200 Q4W | Part 1: 2400 Q4W | Part 1: 1200 Q2W | Part 1: 2400 Q2W | Part 1: 3600 Q2W | Part 1: 3600Q2W + Nivo + Ipi
Number analyzed (Participants) | 16 | 15 | 18 | 12 | 59 | 18 | 12
ug/mL | 142.91 (52.1) | 352.12 (62.7) | 779.90 (43.1) | 325.67 (24.0) | 919.44 (32.8) | 1227.67 (23.3) | 999.60 (29.4)

10. Secondary Outcome: AUC(0-T)-Area Under Curve From Time Zero up to Last Quantifiable Concentration - Part 1
Description: AUC (0-T) represents the observed exposure to a drug (area under the concentration curve) from first exposure until the last quantifiable concentration. Only Part 1 pharmacokinetic evaluable participants were pre-specified to be evaluated in this endpoint.
  1 cycle=28 days for all Arms/Groups except in "Part 1: 3600Q2W + Nivo + Ipi" Arm/Group (1 cycle=42 days)
Time Frame: 0, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96 hours post-dose on Cycle 1 Day 1
Population: All treated participants in Part 1 who have evaluable concentration-time data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | Part 1: 600 Q4W | Part 1: 1200 Q4W | Part 1: 2400 Q4W | Part 1: 1200 Q2W | Part 1: 2400 Q2W | Part 1: 3600 Q2W | Part 1: 3600Q2W + Nivo + Ipi
Number analyzed (Participants) | 16 | 15 | 18 | 12 | 59 | 18 | 12
h*ug/mL | 19594.22 (52.7) | 44821.39 (44.5) | 105171.46 (29.7) | 42835.41 (28.1) | 112123.35 (34.2) | 148321.77 (32.0) | 118041.10 (40.3)

11. Secondary Outcome: AUC(TAU)-Area Under Curve in 1 Dosing Interval - Part 1
Description: Area under the concentration-time curve in 1 dosing interval. Only Part 1 pharmacokinetic evaluable participants were pre-specified to be evaluated in this endpoint.
  1 cycle=28 days for all Arms/Groups except in "Part 1: 3600Q2W + Nivo + Ipi" Arm/Group (1 cycle=42 days)
Time Frame: Cycle 1 Day 1
Population: All treated participants in Part 1 who have evaluable concentration-time data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | Part 1: 600 Q4W | Part 1: 1200 Q4W | Part 1: 2400 Q4W | Part 1: 1200 Q2W | Part 1: 2400 Q2W | Part 1: 3600 Q2W | Part 1: 3600Q2W + Nivo + Ipi
Number analyzed (Participants) | 15 | 14 | 18 | 12 | 56 | 16 | 9
h*ug/mL | 21301.74 (49.5) | 48664.06 (42.9) | 106916.11 (27.3) | 43844.97 (24.8) | 113969.47 (30.8) | 153791.84 (27.9) | 137809.44 (29.5)

12. Secondary Outcome: Observed Serum Concentration at the End of a Dosing Interval (Ctau) - Part 1
Description: BMS-986253 observed serum concentration at the end of a dosing interval (Ctau). Only Part 1 pharmacokinetic evaluable participants were pre-specified to be evaluated in this endpoint.
  1 cycle=28 days for all Arms/Groups except Cycles 1 and 2 (1 cycle=42 days) in "Part 1: 3600Q2W + Nivo + Ipi" Arm/Group
Time Frame: Cycle 1 Day 1
Population: All treated participants in Part 1 who have evaluable concentration-time data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Part 1: 600 Q4W | Part 1: 1200 Q4W | Part 1: 2400 Q4W | Part 1: 1200 Q2W | Part 1: 2400 Q2W | Part 1: 3600 Q2W | Part 1: 3600Q2W + Nivo + Ipi
Number analyzed (Participants) | 15 | 14 | 18 | 12 | 56 | 16 | 9
ug/mL | 6.81 (173.8) | 14.92 (144.4) | 23.68 (692.4) | 55.82 (53.0) | 141.89 (42.6) | 181.84 (46.3) | 175.29 (46.6)

13. Secondary Outcome: Total Body Clearance (CLT) - Part 1
Description: Clearance is the rate of elimination of BMS-986253 from the blood calculated as the rate of elimination divided by serum concentration. Only Part 1 pharmacokinetic evaluable participants were pre-specified to be evaluated in this endpoint.
  1 cycle=28 days for all Arms/Groups except in "Part 1: 3600Q2W + Nivo + Ipi" Arm/Group (1 cycle=42 days)
Time Frame: Cycle 1 Day 1
Population: All treated participants in Part 1 who have evaluable concentration-time data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/h
Arm/Group | Part 1: 600 Q4W | Part 1: 1200 Q4W | Part 1: 2400 Q4W | Part 1: 1200 Q2W | Part 1: 2400 Q2W | Part 1: 3600 Q2W | Part 1: 3600Q2W + Nivo + Ipi
Number analyzed (Participants) | 15 | 14 | 18 | 12 | 56 | 16 | 9
mL/h | 28.17 (49.5) | 24.66 (42.9) | 22.45 (27.3) | 27.37 (24.8) | 21.06 (30.8) | 23.41 (27.9) | 26.12 (29.5)

14. Secondary Outcome: Average Serum Concentration Over a Dosing Interval (Css-avg) - Part 1
Description: BMS-986253 Average concentration over a dosing interval ([AUC(TAU)/tau] (Css-avg) at steady state. Only Part 1 pharmacokinetic evaluable participants were pre-specified to be evaluated in this endpoint.
  1 cycle=28 days for all Arms/Groups except in "Part 1: 3600Q2W + Nivo + Ipi" Arm/Group (1 cycle=42 days)
  Note: C2D1, C3D1, C4D1 were partial samplings only as pre-specified in the protocol and did not include a sampling for each arm.
Time Frame: Cycle 2 Day 1, Cycle 3 Day 1, Cycle 4 Day 1
Population: All treated participants in Part 1 who have evaluable concentration-time data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Part 1: 600 Q4W | Part 1: 1200 Q4W | Part 1: 2400 Q4W | Part 1: 1200 Q2W | Part 1: 2400 Q2W | Part 1: 3600 Q2W | Part 1: 3600Q2W + Nivo + Ipi
Number analyzed (Participants) | 4 | 4 | 8 | 8 | 47 | 13 | 5
ug/mL
  C2D1: number analyzed (Participants) | 0 | 0 | 0 | 8 | 47 | 13 | 5
  C2D1 |  |  |  | 182.48 (26.6) | 487.85 (32.4) | 658.06 (26.2) | 397.96 (32.7)
  C3D1: number analyzed (Participants) | 4 | 4 | 8 | 0 | 0 | 0 | 0
  C3D1 | 59.03 (47.1) | 66.87 (74.2) | 181.94 (19.0) |  |  |  |
  C4D1: number analyzed (Participants) | 0 | 1 | 0 | 3 | 14 | 5 | 0
  C4D1 |  | 115.89 |  | 238.51 (20.1) | 535.44 (37.4) | 590.45 (37.5) |

15. Secondary Outcome: AUC Accumulation Index (AI_AUC) - Part 1
Description: AUC Accumulation Index is defined as the ratio of AUC(TAU) at steady state to AUC(TAU) after the first dose. Only Part 1 pharmacokinetic evaluable participants were pre-specified to be evaluated in this endpoint.
  1 cycle=28 days for all Arms/Groups except in "Part 1: 3600Q2W + Nivo + Ipi" Arm/Group (1 cycle=42 days)
  Note: C2D1, C3D1, C4D1 were partial samplings only as pre-specified in the protocol and did not include a sampling for each arm.
Time Frame: Cycle 2 Day 1, Cycle 3 Day 1, and Cycle 4 Day 1
Population: All treated participants in Part 1 who have evaluable concentration-time data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Part 1: 600 Q4W | Part 1: 1200 Q4W | Part 1: 2400 Q4W | Part 1: 1200 Q2W | Part 1: 2400 Q2W | Part 1: 3600 Q2W | Part 1: 3600Q2W + Nivo + Ipi
Number analyzed (Participants) | 4 | 4 | 8 | 8 | 44 | 10 | 4
Ratio
  C2D1: number analyzed (Participants) | 0 | 0 | 0 | 8 | 44 | 10 | 4
  C2D1 |  |  |  | 1.45 (10.3) | 1.40 (22.8) | 1.34 (20.6) | 1.19 (6.6)
  C3D1: number analyzed (Participants) | 4 | 4 | 8 | 0 | 0 | 0 | 0
  C3D1 | 1.47 (37.4) | 1.07 (16.8) | 1.08 (15.7) |  |  |  |
  C4D1: number analyzed (Participants) | 0 | 1 | 0 | 3 | 12 | 3 | 0
  C4D1 |  | 1.30 |  | 1.77 (20.0) | 1.64 (17.2) | 1.43 (7.1) |

16. Secondary Outcome: Cmax Accumulation Index (AI_Cmax) - Part 1
Description: BMS-986253 Cmax accumulation index (AI_Cmax). Ratio of an exposure measure at steady state to that after the first dose. Only Part 1 pharmacokinetic evaluable participants were pre-specified to be evaluated in this endpoint.
  1 cycle=28 days for all Arms/Groups except in "Part 1: 3600Q2W + Nivo + Ipi" Arm/Group (1 cycle=42 days)
  Note: C2D1, C3D1, C4D1 were partial samplings only as pre-specified in the protocol and did not include a sampling for each arm.
Time Frame: Cycle 2 Day 1, Cycle 3 Day 1, and Cycle 4 Day 1
Population: All treated participants in Part 1 who have evaluable concentration-time data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Part 1: 600 Q4W | Part 1: 1200 Q4W | Part 1: 2400 Q4W | Part 1: 1200 Q2W | Part 1: 2400 Q2W | Part 1: 3600 Q2W | Part 1: 3600Q2W + Nivo + Ipi
Number analyzed (Participants) | 5 | 5 | 9 | 11 | 51 | 14 | 7
Ratio
  C2D1: number analyzed (Participants) | 0 | 0 | 0 | 11 | 51 | 14 | 7
  C2D1 |  |  |  | 1.15 (16.7) | 1.11 (36.5) | 1.21 (18.6) | 1.15 (28.3)
  C3D1: number analyzed (Participants) | 5 | 5 | 9 | 0 | 0 | 0 | 0
  C3D1 | 0.90 (81.6) | 1.05 (16.9) | 0.86 (35.5) |  |  |  |
  C4D1: number analyzed (Participants) | 1 | 1 | 0 | 4 | 21 | 5 | 0
  C4D1 | 1.58 | 1.19 |  | 1.63 (46.0) | 1.36 (26.3) | 0.98 (30.9) |

17. Secondary Outcome: Ctau Accumulation Index (AI_Ctau) - Part 1
Description: Ctau is the observed serum concentration at the end of a dosing interval. Ctau accumulation index (AI_Ctau) is the ratio of an exposure measure at steady state to that after the first dose. Only Part 1 pharmacokinetic evaluable participants were pre-specified to be evaluated in this endpoint. Ctau was reported on non-compartmental analysis day, which is on Cycle 1 Day1, Cycle 2 Day 1, Cycle 3 Day 1, or Cycle 4 Day 1 based on data available.
  1 cycle=28 days for all Arms/Groups except in "Part 1: 3600Q2W + Nivo + Ipi" Arm/Group (1 cycle=42 days)
  Note: C2D1, C3D1, C4D1 were partial samplings only as pre-specified in the protocol and did not include a sampling for each arm.
Time Frame: Cycle 2 Day 1, Cycle 3 Day 1, and Cycle 4 Day 1
Population: All treated participants in Part 1 who have evaluable concentration-time data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Part 1: 600 Q4W | Part 1: 1200 Q4W | Part 1: 2400 Q4W | Part 1: 1200 Q2W | Part 1: 2400 Q2W | Part 1: 3600 Q2W | Part 1: 3600Q2W + Nivo + Ipi
Number analyzed (Participants) | 4 | 4 | 8 | 8 | 44 | 10 | 4
Ratio
  C2D1: number analyzed (Participants) | 0 | 0 | 0 | 8 | 44 | 10 | 4
  C2D1 |  |  |  | 1.90 (22.7) | 1.51 (38.0) | 1.39 (30.7) | 1.10 (21.2)
  C3D1: number analyzed (Participants) | 4 | 4 | 8 | 0 | 0 | 0 | 0
  C3D1 | 1.33 (91.0) | 1.29 (6.5) | 0.90 (53.5) |  |  |  |
  C4D1: number analyzed (Participants) | 0 | 1 | 0 | 3 | 12 | 3 | 0
  C4D1 |  | 1.35 |  | 1.97 (31.5) | 2.01 (35.5) | 1.37 (45.2) |

18. Secondary Outcome: Effective Elimination (T-HALFeff) - Part 1
Description: BMS-986253 effective elimination (T-HALFeff) that explains the degree of accumulation observed for a specific exposure measure. Only Part 1 pharmacokinetic evaluable participants were pre-specified to be evaluated in this endpoint.
  1 cycle=28 days for all Arms/Groups except in "Part 1: 3600Q2W + Nivo + Ipi" Arm/Group (1 cycle=42 days)
  Note: C2D1, C3D1, C4D1 were partial samplings only as pre-specified in the protocol and did not include a sampling for each arm.
Time Frame: Cycle 2 Day 1, Cycle 3 Day 1, and Cycle 4 Day 1
Population: All treated participants in Part 1 who have evaluable concentration-time data
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Part 1: 600 Q4W | Part 1: 1200 Q4W | Part 1: 2400 Q4W | Part 1: 1200 Q2W | Part 1: 2400 Q2W | Part 1: 3600 Q2W | Part 1: 3600Q2W + Nivo + Ipi
Number analyzed (Participants) | 4 | 3 | 6 | 8 | 41 | 9 | 4
Hours
  C2D1: number analyzed (Participants) | 0 | 0 | 0 | 8 | 41 | 9 | 4
  C2D1 |  |  |  | 200.10 (39.12) | 202.89 (76.38) | 185.51 (71.51) | 145.15 (51.41)
  C3D1: number analyzed (Participants) | 4 | 3 | 6 | 0 | 0 | 0 | 0
  C3D1 | 410.31 (275.42) | 222.95 (92.65) | 240.94 (92.57) |  |  |  |
  C4D1: number analyzed (Participants) | 0 | 1 | 0 | 3 | 12 | 3 | 0
  C4D1 |  | 317.87 |  | 283.97 (84.38) | 247.68 (73.44) | 189.42 (22.08) |

19. Secondary Outcome: Time to Maximum Concentration (Tmax) - Part 1
Description: Tmax is defined as the time it takes for a drug to reach the maximum concentration (Cmax) after administration of a drug.
  1 cycle=28 days for all Arms/Groups except in "Part 1: 3600Q2W + Nivo + Ipi" Arm/Group (1 cycle=42 days)
Time Frame: Cycle 1 Day 1
Population: All treated participants in Part 1 who have evaluable concentration-time data
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1: 600 Q4W | Part 1: 1200 Q4W | Part 1: 2400 Q4W | Part 1: 1200 Q2W | Part 1: 2400 Q2W | Part 1: 3600 Q2W | Part 1: 3600Q2W + Nivo + Ipi
Number analyzed (Participants) | 16 | 15 | 18 | 12 | 59 | 18 | 12
Hours | 3.95 [1.0 to 24.0] | 1.00 [0.9 to 4.1] | 3.81 [2.0 to 6.1] | 4.00 [0.9 to 4.2] | 4.00 [1.0 to 23.5] | 2.18 [1.9 to 21.1] | 1.99 [1.9 to 21.8]

20. Secondary Outcome: Serum Trough Concentration (Ctrough) - Part 1
Description: A serum trough concentration (Ctrough) is the concentration reached by a drug immediately before the next dose is administered. Serum trough concentrations (Ctrough) of BMS-986253 will be summarized with descriptive statistics by treatment and visit.
  1 cycle=28 days for all Arms/Groups except in "Part 1: 3600Q2W + Nivo + Ipi" Arm/Group (1 cycle=42 days)
  Note: The timepoints listed were partial samplings only as pre-specified in the protocol and did not include a sampling for each arm.
Time Frame: C1D15, C1D29, C2D1, C2D9, C2D15, C3D1, C4D1, C4D15, C5D1, C7D1, C9D1, C10D1, C14D1, C20D1, and C26D1
Population: All treated participants in Part 1 who have evaluable concentration-time data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 1: 600 Q4W | Part 1: 1200 Q4W | Part 1: 2400 Q4W | Part 1: 1200 Q2W | Part 1: 2400 Q2W | Part 1: 3600 Q2W | Part 1: 3600Q2W + Nivo + Ipi
Number analyzed (Participants) | 10 | 10 | 15 | 11 | 54 | 16 | 11
ng/mL
  C1D15 - Predose: number analyzed (Participants) | 0 | 0 | 0 | 11 | 51 | 14 | 11
  C1D15 - Predose |  |  |  | 59518.0 (49.4) | 149309.4 (37.0) | 221414.7 (26.0) | 166358.6 (43.2)
  C1D29 - Predose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 6
  C1D29 - Predose |  |  |  |  |  |  | 242843.4 (65.2)
  C2D1 - Predose: number analyzed (Participants) | 10 | 10 | 15 | 9 | 54 | 16 | 5
  C2D1 - Predose | 10711.8 (124.6) | 14450.3 (177.5) | 45153.8 (50.4) | 85596.2 (38.1) | 187079.9 (47.5) | 272401.3 (54.1) | 194945.1 (35.3)
  C2D15 - Predose: number analyzed (Participants) | 0 | 0 | 0 | 8 | 46 | 12 | 3
  C2D15 - Predose |  |  |  | 98349.7 (46.0) | 226385.2 (44.5) | 299360.3 (44.3) | 112012.1 (37.6)
  C2D29 - Predose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3
  C2D29 - Predose |  |  |  |  |  |  | 160198.5 (38.2)
  C3D1 - Predose: number analyzed (Participants) | 5 | 6 | 9 | 5 | 27 | 7 | 3
  C3D1 - Predose | 12124.7 (82.5) | 21260.6 (131.9) | 58149.8 (31.5) | 92359.7 (35.7) | 224533.3 (54.9) | 260971.3 (63.9) | 113514.3 (12.4)
  C4D1 - Predose: number analyzed (Participants) | 3 | 3 | 6 | 3 | 23 | 5 | 2
  C4D1 - Predose | 27124.2 (99.1) | 15763.7 (219.2) | 54841.7 (43.6) | 86790.7 (41.8) | 271535.1 (44.9) | 327146.5 (55.7) | 145940.5 (19.8)
  C4D15 - Predose: number analyzed (Participants) | 0 | 0 | 0 | 3 | 14 | 4 | 0
  C4D15 - Predose |  |  |  | 127803.1 (24.5) | 258413.8 (48.1) | 356070.0 (56.9) |
  C5D1 - Predose: number analyzed (Participants) | 0 | 1 | 0 | 3 | 15 | 5 | 0
  C5D1 - Predose |  | 34491.0 |  | 125274.8 (27.4) | 161340.5 (551.8) | 312899.5 (65.2) |
  C7D1 - Predose: number analyzed (Participants) | 1 | 1 | 2 | 0 | 0 | 0 | 0
  C7D1 - Predose | 29506.0 | 51155.0 | 76154.6 (26.5) |  |  |  |
  C9D1 - Predose: number analyzed (Participants) | 0 | 0 | 1 | 3 | 8 | 4 | 0
  C9D1 - Predose |  |  | 48706.0 | 182098.0 (43.0) | 263195.0 (56.6) | 281410.5 (85.2) |
  C10D1 - Predose: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 0
  C10D1 - Predose |  |  | 94273.0 |  |  |  |
  C14D1 - Predose: number analyzed (Participants) | 0 | 1 | 1 | 2 | 4 | 2 | 0
  C14D1 - Predose |  | 95722.0 | 102905.0 | 200795.9 (27.5) | 298491.4 (50.2) | 361774.6 (41.4) |
  C20D1 - Predose: number analyzed (Participants) | 0 | 1 | 1 | 1 | 3 | 1 | 0
  C20D1 - Predose |  | 72607.0 | 116745.0 | 81342.0 | 424725.7 (23.5) | 427000.0 |
  C26D1 - Predose: number analyzed (Participants) | 0 | 1 | 2 | 0 | 0 | 0 | 0
  C26D1 - Predose |  | 56040.0 | 143209.5 (14.8) |  |  |  |

21. Secondary Outcome: Number of Participants With Anti-Drug Antibodies (ADA) - Part 1
Description: Blood samples were evaluated for development of Anti-Drug Antibody (ADA) by a validated electrochemiluminescent (ECL) immunoassay. Baseline is defined as first dose.
  ADA-positive subject: A subject with at least one ADA positive-sample relative to baseline at any time after initiation of treatment.
  Persistent Positive (PP): ADA-positive sample at 2 or more consecutive time points, where the first and last ADA-positive samples are at least 16 weeks apart
  Not PP-Last Sample Positive: Not persistent positive with ADA-positive sample at the last sampling time point
  Other Positive: Not persistent positive but some ADA-positive samples with the last sample being negative
  Neutralizing Positive: At least one ADA-positive sample with neutralizing antibodies detected
  ADA-negative subject: A subject with no ADA-positive sample after the initiation of treatment.
  1 cycle=28 days for all Arms/Groups except in "Part 1: 3600Q2W + Nivo + Ipi" Arm/Group (1 cycle=42 days)
Time Frame: C1D1, C1D2, C1D8, C1D15, C1D22, C2D1, C2D2, C2D8, C2D15, C3D1, C4D1, C4D2, C4D8, C4D15, C4D22, C5D1, C9D1, C14D1, C20D1, C26D1, C32D1, C38D1, 30-day follow-up, 100-day follow-up
Population: All treated participants in Part 1 with baseline and at least one post-baseline evaluable ADA assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: 600 Q4W | Part 1: 1200 Q4W | Part 1: 2400 Q4W | Part 1: 1200 Q2W | Part 1: 2400 Q2W | Part 1: 3600 Q2W | Part 1: 3600Q2W + Nivo + Ipi
Number analyzed (Participants) | 15 | 11 | 16 | 11 | 54 | 15 | 8
Participants
  Baseline ADA positive | 0 | 1 | 0 | 1 | 1 | 0 | 0
  ADA Positive-Overall | 3 | 2 | 4 | 0 | 2 | 0 | 1
  ADA Persistent Positive (PP) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ADA Positive-Not PP last sample positive | 2 | 1 | 1 | 0 | 2 | 0 | 0
  ADA Positive-other positive | 1 | 1 | 3 | 0 | 0 | 0 | 1
  ADA Negative | 12 | 9 | 12 | 11 | 52 | 15 | 7

22. Secondary Outcome: Change From Baseline in Interleukin 8 (IL-8)- Part 1
Description: Change from baseline in IL-8 measured in pg/mL. Baseline is defined as first dose.
  1 cycle=28 days for all Arms/Groups except in "Part 1: 3600Q2W + Nivo + Ipi" Arm/Group (1 cycle=42 days)
  Note: Some timepoints were partial samplings only as pre-specified in the protocol and did not include a sampling for each arm.
Time Frame: C1D2, C1D8, C1D15, C1D22, C1D29, C1D36, C2D1, C2D2, C2D8, C2D15, C2D22, C2D29, C3D1, C3D2, C3D8, C4D1, C4D2, C4D8, C4D15, C4D22, C5D1, C7D1, C8D1, C9D1, C10D1, C11D1, C14D1, C16D1, C17D1, C20D1, C23D1, C26D1, at last dose, and 100 days post last dose
Population: All treated participants in Part 1 with available biomarker data
Measure: Mean (Full Range); unit: pg/mL
Arm/Group | Part 1: 600 Q4W | Part 1: 1200 Q4W | Part 1: 2400 Q4W | Part 1: 1200 Q2W | Part 1: 2400 Q2W | Part 1: 3600 Q2W | Part 1: 3600Q2W + Nivo + Ipi
Number analyzed (Participants) | 16 | 13 | 17 | 12 | 61 | 19 | 12
pg/mL
  Cycle 1 Day 2: number analyzed (Participants) | 16 | 12 | 16 | 11 | 59 | 16 | 12
  Cycle 1 Day 2 | -96.9 [-891.0 to -24.3] | -37.3 [-105.6 to -7.0] | -66.3 [-377.0 to -5.8] | -48.2 [-115.5 to -21.6] | -48.5 [-141.5 to -4.4] | -82.8 [-509.6 to -8.2] | -76.1 [-268.2 to -18.6]
  Cycle 1 Day 8: number analyzed (Participants) | 16 | 12 | 17 | 12 | 61 | 19 | 11
  Cycle 1 Day 8 | -78.2 [-857.0 to -5.0] | -31.4 [-94.0 to -6.2] | -58.6 [-350.0 to -4.8] | -40.3 [-107.0 to -17.2] | -69.8 [-1569.6 to 2.2] | -48.1 [-121.0 to -5.0] | -71.9 [-246.0 to -6.0]
  Cycle 1 Day 15: number analyzed (Participants) | 14 | 13 | 16 | 11 | 58 | 18 | 11
  Cycle 1 Day 15 | -66.2 [-769.0 to 11.0] | -24.4 [-79.0 to 3.0] | -34.3 [-87.0 to -0.3] | -23.6 [-63.0 to -11.0] | -38.0 [-123.2 to 89.0] | -65.8 [-502.5 to -1.0] | -33.5 [-120.0 to -3.0]
  Cycle 1 Day 22: number analyzed (Participants) | 13 | 11 | 15 | 10 | 56 | 17 | 11
  Cycle 1 Day 22 | -48.0 [-561.0 to 24.0] | 17.4 [-30.8 to 277.0] | -41.6 [-240.0 to 11.8] | -33.0 [-77.0 to -18.6] | -71.3 [-1559.0 to 1.7] | -68.1 [-507.2 to -8.2] | -34.3 [-104.0 to -6.0]
  Cycle 1 Day 29: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 10
  Cycle 1 Day 29 |  |  |  |  |  |  | -23.2 [-62.9 to -4.0]
  Cycle 1 Day 36: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 8
  Cycle 1 Day 36 |  |  |  |  |  |  | -29.1 [-66.8 to -10.2]
  Cycle 2 Day 1: number analyzed (Participants) | 10 | 9 | 14 | 10 | 56 | 14 | 9
  Cycle 2 Day 1 | 3.8 [-67.0 to 50.0] | 43.5 [-28.0 to 427.0] | -20.3 [-73.0 to 32.8] | -25.3 [-58.0 to -5.0] | -40.2 [-127.8 to 4.0] | -78.3 [-506.1 to -9.0] | -21.3 [-65.5 to 23.0]
  Cycle 2 Day 2: number analyzed (Participants) | 0 | 0 | 0 | 8 | 46 | 15 | 9
  Cycle 2 Day 2 |  |  |  | -42.5 [-84.0 to -21.6] | -47.3 [-139.4 to 0.0] | -48.2 [-127.1 to -8.2] | -31.5 [-68.6 to -7.7]
  Cycle 2 Day 8: number analyzed (Participants) | 0 | 0 | 0 | 10 | 45 | 15 | 7
  Cycle 2 Day 8 |  |  |  | -35.6 [-77.0 to -18.6] | -44.2 [-136.8 to 0.6] | -77.4 [-508.2 to -8.2] | -26.1 [-68.0 to -5.5]
  Cycle 2 Day 15: number analyzed (Participants) | 7 | 8 | 13 | 10 | 50 | 13 | 6
  Cycle 2 Day 15 | -22.6 [-99.0 to -3.0] | -13.8 [-30.8 to 3.0] | -30.0 [-70.0 to 6.8] | -31.0 [-63.0 to -17.4] | -70.8 [-1569.1 to 3.1] | -74.6 [-501.3 to -7.4] | 9.1 [-22.2 to 56.0]
  Cycle 2 Day 22: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 5
  Cycle 2 Day 22 |  |  |  |  |  |  | -18.7 [-29.4 to -2.8]
  Cycle 2 Day 29: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3
  Cycle 2 Day 29 |  |  |  |  |  |  | -22.7 [-26.9 to -18.0]
  Cycle 3 Day 1: number analyzed (Participants) | 6 | 5 | 10 | 5 | 30 | 9 | 4
  Cycle 3 Day 1 | 2.0 [-82.0 to 44.0] | -4.0 [-25.0 to 30.0] | -16.4 [-49.0 to 21.0] | -25.1 [-38.0 to -8.0] | -86.7 [-1569.6 to 2.3] | -93.5 [-508.2 to -8.1] | -14.4 [-21.0 to 4.0]
  Cycle 3 Day 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Cycle 3 Day 2 |  |  |  |  | -24.9 [-24.9 to -24.9] |  |
  Cycle 3 Day 8: number analyzed (Participants) | 4 | 5 | 8 | 0 | 0 | 0 | 0
  Cycle 3 Day 8 | -36.3 [-113.0 to -7.0] | -24.5 [-34.5 to -15.0] | -37.0 [-77.0 to -13.2] |  |  |  |
  Cycle 3 Day 15: number analyzed (Participants) | 3 | 5 | 8 | 0 | 0 | 0 | 0
  Cycle 3 Day 15 | -44.3 [-117.0 to -2.0] | -20.8 [-31.7 to -14.0] | -24.3 [-46.8 to -5.0] |  |  |  |
  Cycle 3 Day 22: number analyzed (Participants) | 2 | 5 | 6 | 0 | 0 | 0 | 0
  Cycle 3 Day 22 | -53.5 [-107.0 to 0.0] | -15.4 [-27.0 to -2.0] | -16.9 [-43.0 to 23.0] |  |  |  |
  Cycle 4 Day 1: number analyzed (Participants) | 3 | 5 | 6 | 4 | 23 | 6 | 2
  Cycle 4 Day 1 | -30.3 [-101.0 to 18.0] | -8.8 [-26.0 to 13.0] | -15.5 [-28.4 to 3.5] | -18.5 [-38.9 to 1.0] | -102.9 [-1568.8 to 2.0] | -29.6 [-86.0 to 9.0] | -23.8 [-26.4 to -21.1]
  Cycle 4 Day 2: number analyzed (Participants) | 0 | 1 | 0 | 4 | 17 | 5 | 0
  Cycle 4 Day 2 |  | -35.7 [-35.7 to -35.7] |  | -32.0 [-41.7 to -21.3] | -33.5 [-81.6 to 0.5] | -44.0 [-96.9 to -13.6] |
  Cycle 4 Day 8: number analyzed (Participants) | 0 | 1 | 0 | 3 | 15 | 7 | 0
  Cycle 4 Day 8 |  | -32.1 [-32.1 to -32.1] |  | -30.3 [-40.9 to -19.6] | -32.7 [-81.6 to 3.8] | -43.8 [-92.1 to -8.2] |
  Cycle 4 Day 15: number analyzed (Participants) | 0 | 1 | 0 | 3 | 18 | 6 | 0
  Cycle 4 Day 15 |  | -29.0 [-29.0 to -29.0] |  | -26.7 [-38.6 to -17.6] | -34.5 [-122.5 to 6.0] | -46.4 [-90.6 to -8.2] |
  Cycle 4 Day 22: number analyzed (Participants) | 0 | 1 | 0 | 2 | 16 | 6 | 0
  Cycle 4 Day 22 |  | -26.0 [-26.0 to -26.0] |  | -28.8 [-38.5 to -19.1] | -30.6 [-81.1 to 2.7] | -43.8 [-94.5 to -7.6] |
  Cycle 5 Day 1: number analyzed (Participants) | 1 | 0 | 0 | 3 | 16 | 5 | 0
  Cycle 5 Day 1 | 38.0 [38.0 to 38.0] |  |  | -27.3 [-36.0 to -17.7] | -28.2 [-80.3 to 4.9] | -46.8 [-91.7 to -8.2] |
  Cycle 7 Day 1: number analyzed (Participants) | 1 | 2 | 4 | 3 | 10 | 4 | 0
  Cycle 7 Day 1 | -111.0 [-111.0 to -111.0] | -8.0 [-25.0 to 9.0] | -14.6 [-29.7 to -1.7] | -29.3 [-38.5 to -20.0] | -33.0 [-80.8 to -13.6] | -36.9 [-86.6 to -8.2] |
  Cycle 8 Day 1: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Cycle 8 Day 1 |  |  | -21.8 [-21.8 to -21.8] |  |  |  |
  Cycle 9 Day 1: number analyzed (Participants) | 0 | 0 | 1 | 3 | 8 | 2 | 0
  Cycle 9 Day 1 |  |  | -17.0 [-17.0 to -17.0] | -28.2 [-38.5 to -18.6] | -27.8 [-48.3 to -13.6] | -9.1 [-11.0 to -7.1] |
  Cycle 10 Day 1: number analyzed (Participants) | 0 | 0 | 3 | 0 | 0 | 0 | 0
  Cycle 10 Day 1 |  |  | -14.2 [-32.3 to 0.7] |  |  |  |
  Cycle 11 Day 1: number analyzed (Participants) | 0 | 2 | 0 | 3 | 6 | 1 | 0
  Cycle 11 Day 1 |  | -16.0 [-28.0 to -4.0] |  | -30.7 [-37.7 to -21.4] | -24.4 [-39.5 to -13.6] | -7.6 [-7.6 to -7.6] |
  Cycle 14 Day 1: number analyzed (Participants) | 0 | 2 | 1 | 3 | 5 | 0 | 0
  Cycle 14 Day 1 |  | -16.1 [-36.2 to 4.0] | -2.2 [-2.2 to -2.2] | -1.6 [-36.8 to 48.0] | -22.2 [-38.2 to -13.6] |  |
  Cycle 16 Day 1: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Cycle 16 Day 1 |  |  | -1.6 [-1.6 to -1.6] |  |  |  |
  Cycle 17 Day 1: number analyzed (Participants) | 0 | 1 | 2 | 1 | 2 | 0 | 0
  Cycle 17 Day 1 |  | -32.2 [-32.2 to -32.2] | -17.3 [-30.5 to -4.1] | -38.0 [-38.0 to -38.0] | -14.2 [-14.8 to -13.6] |  |
  Cycle 20 Day 1: number analyzed (Participants) | 0 | 1 | 1 | 1 | 3 | 0 | 0
  Cycle 20 Day 1 |  | -30.7 [-30.7 to -30.7] | -32.5 [-32.5 to -32.5] | -34.4 [-34.4 to -34.4] | -17.1 [-23.6 to -13.6] |  |
  Cycle 23 Day 1: number analyzed (Participants) | 0 | 1 | 2 | 0 | 1 | 0 | 0
  Cycle 23 Day 1 |  | -28.9 [-28.9 to -28.9] | -27.1 [-32.2 to -22.0] |  | -22.6 [-22.6 to -22.6] |  |
  Cycle 26 Day 1: number analyzed (Participants) | 0 | 1 | 2 | 0 | 0 | 0 | 0
  Cycle 26 Day 1 |  | -30.8 [-30.8 to -30.8] | -10.0 [-22.6 to 2.5] |  |  |  |
  End of Treatment: number analyzed (Participants) | 2 | 0 | 4 | 5 | 17 | 4 | 2
  End of Treatment | -44.0 [-105.0 to 17.0] |  | -49.5 [-66.0 to -29.0] | -24.6 [-37.0 to -10.0] | -34.5 [-125.0 to 20.0] | -149.1 [-503.2 to -16.0] | -50.9 [-65.0 to -36.8]
  Follow-up 1: number analyzed (Participants) | 0 | 0 | 2 | 0 | 0 | 0 | 0
  Follow-up 1 |  |  | 17.5 [9.0 to 26.0] |  |  |  |

23. Primary Outcome: Objective Response Rate (ORR) - Part 2
Description: Objective Response Rate per blinded independent central review (BICR) is the percentage of participants who have a confirmed complete or partial best overall response (BOR) among participants who have measurable disease at baseline. Complete Response (CR) is defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to =< 10 mm. Partial Response (PR) is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Baseline was defined as evaluations or events that occur before the date and time of the first dose of study treatment or evaluations on the same date and time of the first dose of study treatment were also considered as baseline evaluations. This endpoint was prespecified in the protocol to include only participants in Part 2.
Time Frame: From the date of the first dose to the date of first objectively documented progression per RECIST v1.1 or the date of subsequent therapy, whichever occurred first (up to approximately 22 months)
Population: All randomized participants in Part 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part 2 Arm A: BMS+Nivo+Ipi | Part 2 Arm B: Placebo+Nivo+Ipi
Number analyzed (Participants) | 62 | 60
Percentage of Participants | 14.5 [6.9 to 25.8] | 11.7 [4.8 to 22.6]

24. Secondary Outcome: Progression Free Survival (PFS) - Part 2
Description: Progression free survival (PFS) is defined for all randomized participants as the date from randomization to the date of the documentation of disease progression by BICR or death due to any cause, whichever is earlier.
  Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered progression.
  This endpoint was prespecified in the protocol to include only participants in Part 2.
Time Frame: as for outcome 23
Population: All randomized participants in Part 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 2 Arm A: BMS+Nivo+Ipi | Part 2 Arm B: Placebo+Nivo+Ipi
Number analyzed (Participants) | 62 | 60
Months | 2.103 [1.873 to 3.778] | 3.318 [1.906 to 3.745]
Statistical Analysis 1: Comparison: Part 2 Arm A: BMS+Nivo+Ipi vs Part 2 Arm B: Placebo+Nivo+Ipi; Test type: Other; p = 0.7416, Log Rank; Hazard Ratio, log = 0.94, 95% CI 2-sided [0.61 to 1.45]

25. Secondary Outcome: Number of Participants Experiencing Adverse Events (AEs) - Part 2
Description: An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a pre-existing medical condition in a clinical investigation participant administered study treatment and that does not necessarily have a causal relationship with this treatment. Adverse events are graded on a scale from 1 to 5, with Grade 1 being mild and asymptomatic; Grade 2 is moderate requiring minimal, local or noninvasive intervention; Grade 3 is severe or medically significant but not immediately life-threatening; Grade 4 events are usually severe enough to require hospitalization; Grade 5 events are fatal.
  This endpoint was prespecified in the protocol to include only participants in Part 2.
Time Frame: From first dose up to 100 days after last dose (up to 25 months)
Population: All treated participants in Part 2
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2 Arm A: BMS+Nivo+Ipi | Part 2 Arm B: Placebo+Nivo+Ipi
Number analyzed (Participants) | 62 | 57
Participants | 62 | 56

26. Secondary Outcome: Number of Participants Experiencing Serious Adverse Events (SAEs) - Part 2
Description: A serious adverse event is defined as any untoward medical occurrence that, at any dose: results in death, is life-threatening, requires inpatient hospitalization or causes prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is an important medical event.
Time Frame: From first dose up to 100 days after last dose (up to 25 months)
Population: All treated participants in Part 2
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2 Arm A: BMS+Nivo+Ipi | Part 2 Arm B: Placebo+Nivo+Ipi
Number analyzed (Participants) | 62 | 57
Participants | 44 | 42

27. Secondary Outcome: Number of Participants Experiencing Adverse Events (AEs) Leading to Discontinuation - Part 2
Description: Number of participants with any grade adverse events (AEs) leading to discontinuation of study treatment. An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a pre-existing medical condition in a clinical investigation participant administered study drug and that does not necessarily have a causal relationship with this treatment. Toxicities will be graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.
Time Frame: From first dose up to 100 days after last dose (up to 25 months)
Population: All treated participants in Part 2
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2 Arm A: BMS+Nivo+Ipi | Part 2 Arm B: Placebo+Nivo+Ipi
Number analyzed (Participants) | 62 | 57
Participants | 16 | 23

28. Secondary Outcome: Number of Participants Who Died - Part 2
Description: The number of participants who died due to any cause are summarized.
Time Frame: From first dose up to 100 days after last dose (up to 25 months)
Population: All treated participants in Part 2
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2 Arm A: BMS+Nivo+Ipi | Part 2 Arm B: Placebo+Nivo+Ipi
Number analyzed (Participants) | 62 | 57
Participants | 30 | 17

29. Secondary Outcome: Most Frequently Reported Grade 3 and Grade 4 Laboratory Test Results - Part 2
Description: Laboratory results were graded using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Laboratory tests are graded on a scale from 1 to 5, with Grade 1 being mild and asymptomatic; Grade 2 is moderate requiring minimal, local or noninvasive intervention; Grade 3 is severe or medically significant but not immediately life-threatening; Grade 4 events are usually severe enough to require hospitalization; Grade 5 events are fatal.
  This endpoint was prespecified in the protocol to include only participants in Part 2.
Time Frame: From first dose up to 30 days after last dose (up to 23 months)
Population: All treated participants in Part 2
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2 Arm A: BMS+Nivo+Ipi | Part 2 Arm B: Placebo+Nivo+Ipi
Number analyzed (Participants) | 62 | 57
Participants
  Alanine aminotransferase - Grade 3 | 4 | 6
  Alanine aminotransferase - Grade 4 | 2 | 1
  Aspartate aminotransferase - Grade 3 | 3 | 3
  Aspartate aminotransferase - Grade 4 | 1 | 0
  Phosphate - Grade 3 | 3 | 3
  Sodium - Grade 3 | 6 | 8
  Sodium - Grade 4 | 2 | 0
  Lipase - Grade 3 | 4 | 5
  Lipase - Grade 4 | 5 | 5
  Amylase - Grade 3 | 3 | 4

ADVERSE EVENTS:
Time Frame: Participants were assessed for all-cause mortality from their first dose to their study completion (up to approximately 74 months). SAEs and Other AEs were assessed from first dose to 100 days post the last dose (up to approximately 65 months).
Description: The population for all-cause mortality is all randomized participants. SAEs and Other AEs represents all participants who received at least one dose of study treatment
Arm/Group | Part 1: 600 Q4W | Part 1: 1200 Q4W | Part 1: 2400 Q4W | Part 1: 1200 Q2W | Part 1: 2400 Q2W | Part 1: 3600 Q2W | Part 1: 3600Q2W + Nivo + Ipi | Part 2 Arm A: BMS+Nivo+Ipi | Part 2 Arm B: Placebo+Nivo+Ipi
All-Cause Mortality (participants affected / at risk) | 14/16 | 15/15 | 17/18 | 10/12 | 53/63 | 13/20 | 8/15 | 30/62 | 17/60
Serious Adverse Events (participants affected / at risk) | 13/16 | 10/15 | 13/18 | 7/12 | 31/63 | 12/20 | 9/15 | 44/62 | 42/57
Other Adverse Events (participants affected / at risk) | 16/16 | 14/15 | 18/18 | 11/12 | 59/63 | 19/20 | 15/15 | 61/62 | 54/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: 600 Q4W (N=16) | Part 1: 1200 Q4W (N=15) | Part 1: 2400 Q4W (N=18) | Part 1: 1200 Q2W (N=12) | Part 1: 2400 Q2W (N=63) | Part 1: 3600 Q2W (N=20) | Part 1: 3600Q2W + Nivo + Ipi (N=15) | Part 2 Arm A: BMS+Nivo+Ipi (N=62) | Part 2 Arm B: Placebo+Nivo+Ipi (N=57)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Myocarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Adrenal haemorrhage (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Glucocorticoid deficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypophysitis (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypopituitarism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 4 | 7
Colonic fistula (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 4 | 4
Dysphagia (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastrointestinal vascular malformation haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Immune-mediated enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Rectal prolapse (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Retroperitoneal disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Cardiac death (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Death (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 4 | 1
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 2 | 1
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 3
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hepatorenal syndrome (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1
Bacillus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Kidney infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Lymph gland infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mastitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peritonitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1 | 2 | 1 | 6 | 1 | 0 | 0 | 3
Pneumonia aspiration (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Porphyromonas bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 3 | 1 | 1 | 1 | 1
Urinary tract infection enterococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vascular device infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 3 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
General physical condition abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Troponin T increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 5 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Steroid diabetes (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Spondylitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 4 | 8 | 5 | 17 | 6 | 4 | 6 | 10
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ataxia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Axonal neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Carotid blowout syndrome (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Diabetic coma (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Guillain-Barre syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Middle cerebral artery stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Device occlusion (Product Issues) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Immune-mediated nephritis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 0 | 4 | 0 | 1 | 1 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aortic aneurysm (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Aortic stenosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Superior vena cava syndrome (Vascular disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: 600 Q4W (N=16) | Part 1: 1200 Q4W (N=15) | Part 1: 2400 Q4W (N=18) | Part 1: 1200 Q2W (N=12) | Part 1: 2400 Q2W (N=63) | Part 1: 3600 Q2W (N=20) | Part 1: 3600Q2W + Nivo + Ipi (N=15) | Part 2 Arm A: BMS+Nivo+Ipi (N=62) | Part 2 Arm B: Placebo+Nivo+Ipi (N=57)
Anaemia (Blood and lymphatic system disorders) | 3 | 2 | 5 | 2 | 16 | 7 | 6 | 21 | 14
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 8 | 1
Neutrophilia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Aortic valve incompetence (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 3
Bundle branch block bilateral (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 3 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 4 | 0 | 1 | 0 | 0 | 0 | 2
Deafness (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1
Hypothyroidism (Endocrine disorders) | 1 | 0 | 2 | 0 | 0 | 1 | 2 | 2 | 1
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Vision blurred (Eye disorders) | 2 | 1 | 1 | 0 | 3 | 0 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 4 | 4
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 2 | 1 | 9 | 3 | 3 | 9 | 9
Abdominal pain lower (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 2 | 3 | 3 | 6 | 1
Anorectal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 5 | 6
Constipation (Gastrointestinal disorders) | 3 | 5 | 4 | 1 | 9 | 5 | 1 | 13 | 12
Diarrhoea (Gastrointestinal disorders) | 1 | 3 | 2 | 2 | 14 | 6 | 5 | 27 | 25
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 3 | 1 | 0 | 3 | 4
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 3 | 1 | 0 | 2 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 2 | 1
Epigastric discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1
Gastrointestinal fistula (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal wall thickening (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 5 | 0 | 1 | 3 | 4
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Mucous stools (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 5 | 4 | 4 | 15 | 5 | 3 | 20 | 18
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Oral dysaesthesia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 3 | 0 | 2 | 0 | 1 | 0 | 0
Tongue ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 4 | 2 | 1 | 6 | 2 | 3 | 7 | 9
Asthenia (General disorders) | 2 | 2 | 0 | 2 | 9 | 3 | 2 | 18 | 5
Axillary pain (General disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 1
Chest discomfort (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Chills (General disorders) | 0 | 1 | 0 | 0 | 4 | 2 | 0 | 1 | 5
Face oedema (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Fatigue (General disorders) | 6 | 6 | 6 | 3 | 23 | 9 | 3 | 15 | 22
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Generalised oedema (General disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Influenza like illness (General disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 3
Injection site extravasation (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Localised oedema (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Malaise (General disorders) | 0 | 0 | 1 | 0 | 2 | 2 | 0 | 0 | 0
Medical device pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 1 | 3 | 0 | 0 | 3 | 2
Oedema peripheral (General disorders) | 3 | 0 | 3 | 1 | 3 | 4 | 0 | 4 | 9
Pain (General disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 2 | 0 | 2
Peripheral swelling (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 2 | 3 | 1 | 11 | 5 | 2 | 22 | 16
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 5 | 3
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Seasonal allergy (Immune system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 4 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 5 | 3
Carbuncle (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 3 | 0
Cystitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Herpes zoster reactivation (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Kidney infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 1 | 3 | 0 | 0 | 2 | 0 | 0 | 1
Paronychia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 2 | 0 | 4 | 0 | 1 | 4 | 2
Pneumonia pseudomonal (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Postoperative wound infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 3
Rhinovirus infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sialoadenitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Stoma site infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1 | 0 | 2 | 0 | 2 | 1 | 1
Urinary tract infection (Infections and infestations) | 4 | 2 | 1 | 1 | 7 | 2 | 2 | 3 | 3
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 3 | 2 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Wound secretion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 2 | 1 | 0 | 1 | 4 | 3 | 18 | 13
Amylase increased (Investigations) | 1 | 1 | 2 | 0 | 2 | 1 | 1 | 8 | 4
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 3 | 0 | 3 | 3 | 1 | 15 | 8
Blood albumin decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 7 | 2
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 4 | 0 | 4 | 3 | 0 | 4 | 4
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 6 | 3
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 2
Blood creatinine increased (Investigations) | 0 | 1 | 3 | 2 | 1 | 2 | 0 | 2 | 4
Blood folate decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood iron decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 6
Blood magnesium decreased (Investigations) | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 5 | 1
Blood pH decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood testosterone decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood urea increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 5 | 3
Blood uric acid increased (Investigations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 1 | 0 | 2 | 3 | 3 | 11 | 6
Lipase increased (Investigations) | 1 | 0 | 2 | 1 | 1 | 0 | 2 | 11 | 7
Lymphocyte count decreased (Investigations) | 0 | 0 | 2 | 0 | 2 | 2 | 1 | 4 | 1
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 4 | 2
Platelet count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Protein total decreased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 8 | 4
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 3 | 3 | 0 | 7 | 5 | 1 | 2 | 4
Weight increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 5 | 0 | 4 | 0 | 21 | 3 | 4 | 12 | 12
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 3 | 0 | 1 | 0 | 0 | 0 | 1
Fluid retention (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 7 | 0 | 0 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 2 | 1 | 2 | 13 | 7
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 5 | 0 | 4 | 1 | 1 | 3 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 8 | 3
Hypochloraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 5 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 3 | 0 | 1 | 3 | 0 | 3 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 3 | 0 | 2 | 2 | 0 | 4 | 6
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 2 | 4 | 0 | 6 | 3 | 1 | 8 | 6
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 1 | 3 | 1 | 6 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Iron deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 2 | 1 | 2 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 2 | 1 | 10 | 2 | 1 | 9 | 12
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 4 | 0 | 1 | 7 | 0 | 1 | 6 | 7
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 2
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 1 | 3 | 1 | 1 | 6 | 7
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1 | 8 | 1 | 0 | 7 | 2
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Tendon pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Torticollis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 3
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Central nervous system lesion (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 2 | 1 | 3 | 0 | 0 | 2 | 5
Dysarthria (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 0 | 0 | 2 | 2 | 0 | 2 | 4
Headache (Nervous system disorders) | 1 | 1 | 3 | 0 | 2 | 3 | 1 | 11 | 11
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Hypokinesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 1 | 0 | 0 | 3 | 1 | 0 | 3 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 2
Dysphoria (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hallucination (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 2 | 2 | 0 | 7 | 2 | 1 | 9 | 8
Personality change (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Poor quality sleep (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Cystitis haemorrhagic (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 5 | 1 | 0 | 2 | 3
Hydronephrosis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nocturia (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2
Proteinuria (Renal and urinary disorders) | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Urogenital haemorrhage (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Scrotal oedema (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Scrotal pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2 | 0 | 10 | 1 | 0 | 13 | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 5 | 3 | 3 | 9 | 1 | 2 | 9 | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 2 | 3 | 0 | 2 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 1 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 2 | 1
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 2 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 2 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 0 | 2 | 0 | 0 | 1 | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 4 | 0 | 0 | 2 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Nail bed bleeding (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nail ridging (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 3
Panniculitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 12 | 2 | 1 | 18 | 18
Rash (Skin and subcutaneous tissue disorders) | 1 | 3 | 1 | 0 | 5 | 0 | 2 | 10 | 10
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 1 | 1 | 0 | 2 | 7 | 11
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Vitiligo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 5 | 2
Embolism (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Hot flush (Vascular disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 2 | 4 | 1 | 3 | 0 | 0 | 3 | 3
Hypotension (Vascular disorders) | 0 | 1 | 1 | 1 | 1 | 2 | 1 | 0 | 3
Lymphoedema (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Superior vena cava syndrome (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-17): https://cdn.clinicaltrials.gov/large-docs/32/NCT03400332/Prot_SAP_000.pdf